CLINICAL TRIAL: NCT03367819
Title: A Phase 1/2 Open-label, Multi-center, Safety, Preliminary Efficacy and Pharmacokinetic (PK) Study of Isatuximab (SAR650984) in Combination With REGN2810, or Isatuximab Alone, in Patients With Advanced Malignancies
Brief Title: Isatuximab in Combination With REGN2810 (Cemiplimab) in Patients With Advanced Malignancies
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: The study was stopped after interim analysis indicated that overall result was not sufficient to satisfy per-protocol criteria to move forward in metastatic, castration-resistant prostate cancer (mCRPC) and non-small cell lung cancer (NSCLC) cohorts.
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ACT15319; 2017-002846-61 (EudraCT Number); U1111-1197-7792 (Registry Identifier: ICTRP)
Record Dates: First submitted 2017-12-05; First posted 2017-12-11 (Actual); Results first posted 2022-05-16 (Actual); Last update posted 2022-05-16 (Actual); Status verified 2022-04

CONDITIONS: Prostate Cancer; Non-small Cell Lung Cancer
Keywords: Anti-CD38 monoclonal antibody
MeSH Terms: conditions — Prostatic Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — isatuximab; cemiplimab

STUDY DESIGN:
Intervention Model Description: Random assignment used only for allocation to Cohort A-1 or A-2
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Phase 1: mCRPC/NSCLC (Experimental): Isatuximab dose 1 and REGN2810 predefined dose
  Interventions: Drug: Isatuximab SAR650984; Drug: Cemiplimab REGN2810
- Cohort A-1: mCRPC, isatuximab and REGN2810 combination (Experimental): Participants with mCRPC will be given isatuximab dose determined in Phase 1 arm of study and REGN2810 predefined dose
  Interventions: Drug: Isatuximab SAR650984; Drug: Cemiplimab REGN2810
- Cohort A-2: mCRPC, isatuximab monotherapy (Experimental): Participants with mCRPC will be given isatuximab dose 2
  Interventions: Drug: Isatuximab SAR650984
- Phase 2 Cohort B: NSCLC (Experimental): Participants with NSCLC will be given isatuximab dose determined in Phase 1 arm of study and REGN2810 predefined dose
  Interventions: Drug: Isatuximab SAR650984; Drug: Cemiplimab REGN2810
- Possibly Phase 2 Cohort C: mCRPC (Experimental): Isatuximab dose 3 will be given in combination with REGN2810 predefined dose or isatuximab dose 3 will be given as monotherapy in participants with mCRPC
  Interventions: Drug: Isatuximab SAR650984; Drug: Cemiplimab REGN2810
- Possibly Phase 2 Cohort D: NSCLC (Experimental): Isatuximab dose 3 will be given in combination with REGN2810 predefined dose
  Interventions: Drug: Isatuximab SAR650984; Drug: Cemiplimab REGN2810

INTERVENTIONS:
Drug: Isatuximab SAR650984 — Pharmaceutical form: solution for infusion
  Route of administration: intravenous
  Other Names: Sarclisa
Drug: Cemiplimab REGN2810 — Pharmaceutical form: solution for infusion
  Route of administration: intravenous
  Arms: Cohort A-1: mCRPC, isatuximab and REGN2810 combination; Phase 1: mCRPC/NSCLC; Phase 2 Cohort B: NSCLC; Possibly Phase 2 Cohort C: mCRPC; Possibly Phase 2 Cohort D: NSCLC

SUMMARY:
Primary Objectives:

* To characterize the safety and tolerability of isatuximab in combination with REGN2810 in participants with metastatic, castration-resistant prostate cancer (mCRPC) who were naïve to anti-programmed cell death-1 (PD-1)/programmed cell death-ligand 1 (PD-L1)-containing therapy, or non-small cell lung cancer (NSCLC) who progressed on anti-PD-1/PD-L1-containing therapy, and to confirm the recommended Phase 2 dose (RP2D).
* To assess the response rate of isatuximab in combination with REGN2810 in participants with either mCRPC who were anti-PD-1/PD-L1 therapy naive, or NSCLC who progressed on anti-PD-1/PD-L1 therapy, or of isatuximab as single agent in participants with mCRPC.

Secondary Objectives:

* To evaluate the safety of the combination of isatuximab with REGN2810 or isatuximab monotherapy.
* To evaluate the immunogenicity of isatuximab and REGN2810.
* To characterize the pharmacokinetic (PK) profile of isatuximab single agent or in combination with REGN2810, and to characterize the PK of REGN2810 in combination with isatuximab.
* To assess overall efficacy of isatuximab in combination with REGN2810 or as a single agent.

DETAILED DESCRIPTION:
The total study duration per participant was up to 28 months including an up to 28 days screening period, an up to 24 months treatment period, and a 3 months safety follow up period.

ELIGIBILITY:
Inclusion Criteria:

* Participants must had a known diagnosis of either metastatic castration-resistant prostate cancer (mCRPC) or non-small cell lung cancer (NSCLC) with evidence of measurable disease.
* Failure of, inability to, or refusal to receive standard of care.
* Greater than or equal to (>=) 18 years of age.

Exclusion Criteria:

* Prior exposure to isatuximab or participation in clinical studies with isatuximab.
* For participants with mCRPC, prior exposure to any agent (approved or investigational) that blocks the PD-1/PD-L1 pathway.
* Evidence of other immune related disease /conditions.
* History of non-infectious pneumonitis requiring steroids or current pneumonitis; history of the thoracic radiation.
* Had received a live-virus vaccination within 28 days of planned treatment start. Seasonal flu vaccines that do not contain live virus were permitted.
* Prior solid organ or hematologic transplant.
* Eastern Cooperative Oncology Group performance status (PS) >=2.
* Poor bone marrow reserve.
* Poor organ function.

The above information was not intended to contain all considerations relevant to a participant's potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2018-01-04 (Actual); Primary Completion 2021-03-10 (Actual); Study Completion 2021-03-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (16):
- United States (5):
  - Investigational Site Number 8400003, Birmingham, Alabama
  - Investigational Site Number 8400007, Atlanta, Georgia
  - Investigational Site Number 8400002, Hackensack, New Jersey
  - Investigational Site Number 8400005, Nashville, Tennessee
  - Investigational Site Number 8400004, Houston, Texas
- France (2):
  - Investigational Site Number 2500002, Bordeaux
  - Investigational Site Number 2500001, Villejuif
- Italy (5):
  - Investigational Site Number 3800003, Rozzano, Milano
  - Investigational Site Number 3800001, Orbassano, Torino
  - Investigational Site Number 3800006, Napoli
  - Investigational Site Number 3800004, Padua
  - Investigational Site Number 3800005, Verona
- Taiwan (2):
  - Investigational Site Number 1580002, Tainan
  - Investigational Site Number 1580001, Taipei
- United Kingdom (2):
  - Investigational Site Number 8260001, Sutton, Surrey
  - Investigational Site Number 8260002, Newcastle upon Tyne

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- [Derived] Zucali PA, Lin CC, Carthon BC, Bauer TM, Tucci M, Italiano A, Iacovelli R, Su WC, Massard C, Saleh M, Daniele G, Greystoke A, Gutierrez M, Pant S, Shen YC, Perrino M, Meng R, Abbadessa G, Lee H, Dong Y, Chiron M, Wang R, Loumagne L, Lepine L, de Bono J. Targeting CD38 and PD-1 with isatuximab plus cemiplimab in patients with advanced solid malignancies: results from a phase I/II open-label, multicenter study. J Immunother Cancer. 2022 Jan;10(1):e003697. doi: 10.1136/jitc-2021-003697. PMID 35058326

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study was conducted at 16 active sites in 5 countries. A total of 44 participants were enrolled between 04 January 2018 and 18 January 2019 and received isatuximab in combination with REGN2810.
Pre-assignment Details: The study was planned to be conducted in 3 parts: Phase 1 part (safety run-in), Phase 2 part (efficacy) and Cross-over part (a subpart of Cohort A-2). Since the enrolled participants (24 for metastatic, castration-resistant prostate cancer [mCRPC] Cohort A-1 and 20 participants for non-small cell lung cancer [NSCLC] Cohort B) did not achieve the pre-defined efficacy criteria, the study was stopped per-protocol and thus, few planned outcome measures were not analyzed.
Groups:
- mCRPC: Isatuximab + REGN2810: Participants with mCRPC received intravenous (IV) infusion of isatuximab 10 milligrams per kilogram (mg/kg) once weekly (QW) for 3 weeks (i.e., on Days 1, 8 and 15) of Cycle 1 and then on Day 1 of Cycle 2 and subsequent cycles (each cycle of 21 days), along with REGN2810 350 mg IV infusion on Day 1 of each 21-day treatment Cycle (maximum duration: up to 2 years).
- NSCLC: Isatuximab + REGN2810: Participants with NSCLC received IV infusion of isatuximab 10 mg/kg QW for 3 weeks (i.e., on Days 1, 8 and 15) of Cycle 1 and then on Day 1 of Cycle 2 and subsequent cycles (each cycle of 21 days), along with REGN2810 350 mg IV infusion on Day 1 of each 21-day treatment Cycle (maximum duration: up to 2 years).
Period: Overall Study
Arm/Group | mCRPC: Isatuximab + REGN2810 | NSCLC: Isatuximab + REGN2810
Started | 24 | 20
Completed | 0 | 1
Not Completed | 24 | 19
Not completed — Adverse Event | 4 | 4
Not completed — Progressive Disease | 15 | 13
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Other | 4 | 2

BASELINE CHARACTERISTICS:
Population: Analysis was performed on all-treated population which included all participants who signed the study informed consent (IC) and received at least 1 dose (even incomplete) of the study treatments, either isatuximab or REGN2810.
Arm/Group | mCRPC: Isatuximab + REGN2810 | NSCLC: Isatuximab + REGN2810 | Total Title
Number analyzed (Participants) | 24 | 20 | 44
Age, Continuous [Mean (Standard Deviation); unit: years] | 70.7 (6.5) | 65.4 (5.8) | 68.3 (6.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 6 | 6
  Male | 24 | 14 | 38
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 6 | 5 | 11
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 18 | 10 | 28
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 4 | 4

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Dose Limiting Toxicities (DLTs)
Description: DLTs: adverse events occurring during 1st treatment cycle, unless due to disease progression/to cause obviously unrelated to investigational medicinal product (IMP) which included:hematological abnormalities: Grade(G) 4 neutropenia(N) for 7/more consecutive days, G3 to G4 N with fever (temperature greater than or equal to [>=] 38.5 degree Celsius on more than 1 occasion) or microbiologically/radiographically documented infection, G3 to G4 thrombocytopenia with clinically significant bleeding. Non-hematological abnormalities: G4 non-hematologic AE, G>=2 uveitis, G3 non-hematological AE lasting greater than (>)3 days (except G3 fatigue, allergic reaction/hypersensitivity attributed to isatuximab or REGN2810 and G3 or G4 clinically non-significant laboratory abnormality), delay in initiation of Cycle 2 >14 days due to treatment related laboratory abnormalities/AE. Any other toxicity that Investigator and Sponsor deemed to be dose-limiting, regardless of grade, was also considered as DLT.
Time Frame: Cycle 1 (21 days)
Population: Analysis was performed on DLT evaluable population which included participants who received the planned doses of isatuximab and REGN2810 during Cycle 1, and who completed the DLT observation period after the first IMP administration, unless they discontinued the study treatment(s) due to DLT.
Measure: Count of Participants; unit: Participants
Arm/Group | mCRPC: Isatuximab + REGN2810 | NSCLC: Isatuximab + REGN2810
Number analyzed (Participants) | 5 | 1
Participants | 0 | 0

2. Primary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs) and Treatment-emergent Serious Adverse Events (TESAEs)
Description: An AE was defined as any untoward medical occurrence in a participant who received study drug and did not necessarily have to have a causal relationship with the treatment. Serious adverse events (SAEs) was any untoward medical occurrence that at any dose: resulted in death, was life-threatening, required inpatient hospitalization or prolongation of existing hospitalization, resulted in persistent or significant disability/incapacity, was a congenital anomaly/birth defect, was a medically important event. TEAEs were defined as AEs that developed, worsened or became serious during the TEAE period (defined as the time from the first dose of study treatment up to 30 days after the last dose of study treatment). TEAEs included both SAEs and non-SAEs.
Time Frame: From Baseline up to 30 days after the last dose of study treatments (maximum duration: up to 2 years)
Population: Analysis was performed on all-treated population.
Measure: Count of Participants; unit: Participants
Arm/Group | mCRPC: Isatuximab + REGN2810 | NSCLC: Isatuximab + REGN2810
Number analyzed (Participants) | 24 | 20
Participants
  Any TEAEs | 24 | 20
  Any TESAEs | 11 | 14

3. Primary Outcome: Number of Participants With Laboratory Abnormalities: Hematological Parameters
Description: Hematological parameters assessed were anemia, white blood cell (WBC) decreased, platelet count decreased, lymphocyte count decreased and neutrophil count decreased. Abnormality criteria was based on National Cancer Institute Common Terminology Criteria for Adverse Event version 4.03 (NCI-CTCAE v 4.03), where Grade 1 = Mild; Grade 2 = Moderate; Grade 3 = Severe; Grade 4 = Potentially Life Threatening. Only those categories in which at least 1 participant had data were reported.
Time Frame: From Baseline up to 30 days after the last dose of study treatments (maximum duration: up to 2 years)
Population: Analysis was performed on all-treated population. Here, overall number of participants analyzed = participants evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | mCRPC: Isatuximab + REGN2810 | NSCLC: Isatuximab + REGN2810
Number analyzed (Participants) | 23 | 20
Participants
  Anemia: Grade 1 | 10 | 9
  Anemia: Grade 2 | 9 | 2
  Anemia: Grade 3 | 4 | 3
  WBC decreased: Grade 1 | 8 | 2
  WBC decreased: Grade 2 | 5 | 0
  Platelet count decreased: Grade 1 | 5 | 1
  Platelet count decreased: Grade 2 | 2 | 0
  Platelet count decreased: Grade 3 | 1 | 0
  Lymphocyte count decreased: Grade 1 | 4 | 7
  Lymphocyte count decreased: Grade 2 | 8 | 4
  Lymphocyte count decreased: Grade 3 | 5 | 2
  Lymphocyte count decreased: Grade 4 | 1 | 0
  Neutrophil count decreased: Grade 1 | 3 | 2
  Neutrophil count decreased: Grade 2 | 2 | 0

4. Primary Outcome: Number of Participants With Laboratory Abnormalities: Electrolytes
Description: Abnormal electrolytes parameters assessed were hyponatremia, hypokalemia, hyperkalemia, hypocalcemia, hypercalcemia, hypoalbuminemia and hyperglycemia. Abnormality criteria was based on NCI-CTCAE v 4.03, where Grade 1 = Mild; Grade 2 = Moderate; Grade 3 = Severe; Grade 4 = Potentially Life Threatening. Only those categories in which at least 1 participant had data were reported.
Time Frame: From Baseline up to 30 days after the last dose of study treatments (maximum duration: up to 2 years)
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | mCRPC: Isatuximab + REGN2810 | NSCLC: Isatuximab + REGN2810
Number analyzed (Participants) | 23 | 20
Participants
  Hyponatremia: Grade 1 | 8 | 8
  Hypokalemia: Grade 1 | 3 | 2
  Hyperkalemia: Grade 1 | 3 | 2
  Hypocalcemia: Grade 1 | 6 | 3
  Hypocalcemia: Grade 2 | 1 | 0
  Hypercalcemia: Grade 1 | 1 | 1
  Hypercalcemia: Grade 2 | 0 | 1
  Hypoalbuminemia: Grade 1 | 6 | 2
  Hypoalbuminemia: Grade 2 | 1 | 3
  Hypoalbuminemia: Grade 3 | 0 | 1
  Hyperglycemia: Grade 1 | 11 | 3
  Hyperglycemia: Grade 2 | 5 | 5
  Hyperglycemia: Grade 3 | 1 | 0
  Hypoglycemia: Grade 1 | 0 | 1
  Hypoglycemia: Grade 2 | 0 | 1

5. Primary Outcome: Number of Participants With Laboratory Abnormalities: Renal Parameters
Description: Abnormal renal parameters assessed were creatinine clearance (CrCl), creatinine increased and hyperuricemia. Creatinine clearance was assessed in categories: >=60 - less than (<) 90 milliliters per minute per 1.73 square meter (mL/min/1.73m^2), >=30 - <60 mL/min/1.73m^2, >=15 - <30 mL/min/1.73m^2 and <15 mL/min/1.73m^2. Creatinine increased and hyperuricemia abnormality criteria was based on NCI-CTCAE v 4.03, where Grade 1 = Mild; Grade 2 = Moderate; Grade 3 = Severe; Grade 4 = Potentially Life Threatening. For all these 3 parameters, only those categories in which at least 1 participant had data were reported.
Time Frame: From Baseline up to 30 days after the last dose of study treatments (maximum duration: up to 2 years)
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | mCRPC: Isatuximab + REGN2810 | NSCLC: Isatuximab + REGN2810
Number analyzed (Participants) | 23 | 20
Participants
  CrCl: >=60 - <90 mL/min/1.73m^2 | 6 | 13
  CrCl: >=30 - <60 mL/min/1.73m^2 | 11 | 2
  Creatinine increased: Grade 1 | 18 | 15
  Hyperuricemia: Grade 3 | 2 | 3
  Hyperuricemia: Grade 4 | 1 | 0

6. Primary Outcome: Number of Participants With Laboratory Abnormalities: Liver Function Parameters
Description: Abnormal liver function parameters assessed were aspartate aminotransferase (AST) increased, alanine aminotransferase (ALT) increased, alkaline phosphatase (ALP) increased, blood bilirubin (BB) increased. Abnormality criteria was based on NCI-CTCAE v 4.03, where Grade 1 = Mild; Grade 2 = Moderate; Grade 3 = Severe; Grade 4 = Potentially Life Threatening. Only those categories in which at least 1 participant had data were reported.
Time Frame: From Baseline up to 30 days after the last dose of study treatments (maximum duration: up to 2 years)
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | mCRPC: Isatuximab + REGN2810 | NSCLC: Isatuximab + REGN2810
Number analyzed (Participants) | 23 | 20
Participants
  AST increased: Grade 1 | 6 | 2
  AST increased: Grade 2 | 1 | 0
  ALT increased: Grade 1 | 2 | 0
  ALP increased: Grade 1 | 3 | 9
  ALP increased: Grade 2 | 4 | 0
  ALP increased: Grade 3 | 6 | 0
  BB increased: Grade 1 | 2 | 1

7. Primary Outcome: Overall Response Rate (ORR): Percentage of Participants With Overall Response
Description: For participants with mCRPC, response was defined as achieving complete response (CR) or partial response (PR) as best overall response (BOR) for soft tissue assessed and confirmed by the Investigators and/or a prostate-specific antigen (PSA) decline of >=50 percent (%) from Baseline that was subsequently confirmed per Prostate Cancer Clinical Trials Working Group 3 (PCWG3) criteria. For participants with NSCLC, ORR was defined as the percentage of participants with CR or PR as BOR according to RECIST 1.1. criteria. Per RECIST 1.1. criteria, CR: disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must had reduction in short axis to <10 millimeters (mm) and PR: at least a 30% decrease in the sum of diameters of target lesions, taking as reference the Baseline sum diameters.
Time Frame: From the date of randomization to the date of first documentation of progression or death due to any cause, whichever occurred first (maximum duration: up to 2 years)
Population: Analysis was performed on all-treated population.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | mCRPC: Isatuximab + REGN2810 | NSCLC: Isatuximab + REGN2810
Number analyzed (Participants) | 24 | 20
percentage of participants | 4.2 [0.2 to 18.3] | 0 [0.0 to 13.9]

8. Secondary Outcome: Number of Participants With Anti-drug Antibodies (ADA) Response Against Isatuximab, Post Treatment
Description: ADA response were categorized as treatment boosted ADA and treatment-induced ADA. Treatment boosted ADA was defined as pre-existing ADAs with a significant increase in the ADA titer during the study compared to the Baseline titer. Treatment-induced ADA was defined as ADA that developed at any time during the ADA on-study observation period in participants without pre-existing ADA (including participants without pretreatment samples).
Time Frame: From Baseline up to 2 years
Population: Analyzed on ADA population: all participants who signed the study IC and received at least 1 dose (even incomplete) of the study treatments, either isatuximab or REGN2810 and had at least 1 ADA non-missing results after the first dose of study treatment. Here, 'overall number of participants analyzed'= participants evaluable for this outcome measure. For this outcome measure, combined ADA analysis was planned and performed for participants with mCRPC and NSCLC.
Measure: Count of Participants; unit: Participants
Groups:
- mCRPC + NSCLC : Isatuximab + REGN2810: Participants with mCRPC and NSCLC received IV infusion of isatuximab 10 mg/kg QW for 3 weeks (i.e., on Days 1, 8 and 15 of Cycle 1) and then on Day 1 of Cycle 2 and subsequent cycles (each cycle of 21 days), along with REGN2810 350 mg IV infusion on Day 1 of each 21-day treatment Cycle (maximum duration: up to 2 years).
Arm/Group | mCRPC + NSCLC : Isatuximab + REGN2810
Number analyzed (Participants) | 39
Participants | 0

9. Secondary Outcome: Number of Participants With Anti-drug Antibodies (ADA) Response Against REGN2810, Post Treatment
Description: as for outcome 8
Time Frame: From Baseline up to 2 years
Population: Analysis was performed on ADA population. Here, 'overall number of participants analyzed' = participants evaluable for this outcome measure. For this outcome measure, combined ADA analysis was planned and performed for participants with mCRPC and NSCLC.
Measure: Count of Participants; unit: Participants
Arm/Group | mCRPC + NSCLC : Isatuximab + REGN2810
Number analyzed (Participants) | 39
Participants | 1

10. Secondary Outcome: Pharmacokinetics (PK): Maximum Observed Plasma Concentration (Cmax) After the First Infusion of Isatuximab
Description: Cmax was defined as the maximum observed plasma concentration. Cmax analysis was done separately for isatuximab for participants with mCRPC and NSCLC.
Time Frame: At start of infusion (SOI), before actual end of infusion (EOI), EOI+4 hours, 72 hours and 168 hours post-dose on Day 1 of Cycle 1
Population: Analyzed on PK population which included all participants who signed the study IC and received at least 1 dose (even incomplete) of the study treatments, either isatuximab or REGN2810 and had at least 1 drug concentration after the first dose of study treatment. Here, overall number of participants analyzed = participants with available data for this outcome measure.
Measure: Mean (Standard Deviation); unit: micrograms per milliliter
Groups:
- mCRPC: Isatuximab: Participants with mCRPC received IV infusion of isatuximab 10 mg/kg QW for 3 weeks (i.e., on Days 1, 8 and 15 of Cycle 1) and then on Day 1 of Cycle 2 and subsequent cycles (each cycle of 21 days) (Maximum duration: up to 2 years).
- NSCLC: Isatuximab: Participants with NSCLC received IV infusion of isatuximab 10 mg/kg QW for 3 weeks (i.e., on Days 1, 8 and 15 of Cycle 1) and then on Day 1 of Cycle 2 and subsequent cycles (each cycle of 21 days)) (Maximum duration: up to 2 years).
Arm/Group | mCRPC: Isatuximab | NSCLC: Isatuximab
Number analyzed (Participants) | 17 | 16
micrograms per milliliter | 291 (67.9) | 280 (54.5)

11. Secondary Outcome: Pharmacokinetics (PK): Maximum Observed Plasma Concentration (Cmax) After the First Infusion of REGN2810
Description: Cmax was defined as the maximum observed plasma concentration. Cmax analysis was done separately for REGN2810 for participants with mCRPC and NSCLC.
Time Frame: At SOI, before actual EOI, EOI+4 hours, 72 hours, 168 hours, and 336 hours post-dose on Day 1 of Cycle 1
Population: Analysis was performed on PK population. Here, overall number of participants analyzed = participants with available data for this outcome measure.
Measure: Mean (Standard Deviation); unit: milligrams per liter
Groups:
- mCRPC: REGN2810: Participants with mCRPC received IV infusion of REGN2810 350 mg IV infusion on Day 1 of each 21-day treatment Cycle (Maximum duration: up to 2 years).
- NSCLC: REGN2810: Participants with NSCLC received IV infusion of REGN2810 350 mg IV infusion on Day 1 of each 21-day treatment Cycle (Maximum duration: up to 2 years).
Arm/Group | mCRPC: REGN2810 | NSCLC: REGN2810
Number analyzed (Participants) | 19 | 17
milligrams per liter | 102 (26.1) | 116 (21.4)

12. Secondary Outcome: Pharmacokinetics: Area Under the Plasma Concentration Versus Time Curve From Time 0 to 168 Hours (AUC0-168 hr) After the First Administration of Isatuximab
Description: AUC0-168 hr was defined as the area under the plasma concentration-time curve from time zero to 168h and was calculated using the trapezoidal method over the dosing interval (i.e., 7 days) for isatuximab alone.
Time Frame: At SOI, before actual EOI, EOI+4 hours, 72 hours and 168 hours post-dose on Day 1 of Cycle 1
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: micrograms*hour per milliliter
Arm/Group | mCRPC: Isatuximab | NSCLC: Isatuximab
Number analyzed (Participants) | 16 | 14
micrograms*hour per milliliter | 28400 (6610) | 24500 (5510)

13. Secondary Outcome: Pharmacokinetics: Area Under the Plasma Concentration Versus Time Curve From Time 0 to 504 Hours (AUC0-504 hr) After the First Administration of REGN2810
Description: AUC0-504 hr was defined as the area under the plasma concentration-time curve from time zero to 504h and was calculated using the trapezoidal method over the dosing interval (i.e., 21 days) for REGN2810 alone.
Time Frame: At SOI, before actual EOI, EOI+4 hours, 72 hours, 168 hours, 336 hours and 504 hours post-dose on Day 1 of Cycle 1
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: milligrams*day per liter
Arm/Group | mCRPC: REGN2810 | NSCLC: REGN2810
Number analyzed (Participants) | 19 | 7
milligrams*day per liter | 903 (257) | 1020 (229)

14. Secondary Outcome: Best Percent-change From Baseline in Tumor Burden
Description: Tumor burden change was defined as the best percent-change from Baseline in a sum of the diameters (longest for non-nodal lesion, short axis for nodal lesions) for all target lesions.
Time Frame: Up to 2 years
Population: Analysis was performed on all-treated population.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | mCRPC: Isatuximab + REGN2810 | NSCLC: Isatuximab + REGN2810
Number analyzed (Participants) | 24 | 20
percent change | 12.9 (47.6) | 0.7 (10.1)

15. Secondary Outcome: Duration of Response (DOR)
Description: DOR: defined as time (in months) from date of first response (PR or CR in radiographic objective response, or PSA decline >=50% for participants with mCRPC) that was subsequently confirmed to the date of first disease progression (PD) or death, whichever occurred first. PD included radiographic disease progression or unequivocal clinical progression. RECIST 1.1 criteria was used to assess radiographic PD in participants with NSCLC and PCWG3 criteria for participants with mCRPC. Per RECIST 1.1 criteria, CR: disappearance of all target lesions. Any pathological lymph nodes (whether target/non-target) must had reduction in short axis to <10 mm and PR: at least a 30% decrease in sum of diameters of target lesions, taking as reference baseline sum diameters. PD: at least a 20% increase in sum of diameters of target lesions, taking as reference smallest sum on study (Baseline sum if that was smallest), sum with an absolute increase of at least 5 mm and appearance of 1 or more new lesions.
Time Frame: From the date of first response until disease progression or death, whichever occurred first (maximum duration: up to 2 years)
Population: Analysis was performed on subset of participants who had response. Here, '0' in 'overall number of participants analyzed represents that DOR could only be analyzed in participants who achieved a response. As no participant in the NSCLC cohort achieved any response, no DOR is available.
Measure: Mean (Standard Deviation); unit: months
Arm/Group | mCRPC: Isatuximab + REGN2810 | NSCLC: Isatuximab + REGN2810
Number analyzed (Participants) | 1 | 0
months | 4.17 |

16. Secondary Outcome: Progression-free Survival (PFS)
Description: For mCRPC participants, PFS was defined as the time (in months) from first study treatment administration to the date of first documented disease progression or the date of death from any cause, whichever occurred first. Disease progression included radiographic disease progression (per PCWG3 criteria) or unequivocal clinical progression. For NSCLC participants, PFS was defined as the time from first study treatment administration to the date of first documented radiographic progression (PD) (per RECIST 1.1) or the date of death from any cause, whichever occurred first. Per RECIST 1.1 criteria, PD was defined as at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (this included the Baseline sum if that is the smallest on study). The sum must also demonstrate an absolute increase of at least 5 mm. Appearance of 1 or more new lesions was also considered as progression. Analysis was performed using Kaplan-Meier method.
Time Frame: From the date of the first study treatment administration to the date of first documented disease progression or death of any cause, whichever occurred first (maximum duration: up to 2 years)
Population: Analysis was performed on all-treated population.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | mCRPC: Isatuximab + REGN2810 | NSCLC: Isatuximab + REGN2810
Number analyzed (Participants) | 24 | 20
months | 2.30 [1.906 to 4.271] | 4.01 [1.938 to 4.074]

17. Secondary Outcome: Percentage of Participants With Disease Control (DC) >=6 Months
Description: Disease control: defined as percentage of participants with confirmed CR/PR/stable disease (SD), as assessed by Investigator PCWG3 modified RECIST 1.1 criteria relative to total number of participants in analysis population. Per PCWG3 modified RECIST 1.1 criteria, CR: disappearance of all target lesions. Any pathological lymph nodes (whether target/non-target) must had reduction in short axis to <10 mm, PR: at least a 30% decrease in sum of diameters of target lesions, taking as reference Baseline sum diameters and SD: neither sufficient shrinkage from the Baseline to qualify for PR nor sufficient increase to qualify for PD, taking as reference smallest sum diameters while on study. PD: at least a 20% increase in sum of diameters of target lesions, taking as reference smallest sum on study, sum with an absolute increase of diameter of at least 5 mm and appearance of 1 or more new lesions.
Time Frame: From the date of first response to the date of first documented disease progression or death (due to any cause) (maximum duration: up to 2 years)
Population: Analysis was performed on all-treated population. Here, '0' in 'overall number of participants analyzed represents that data for this outcome measure was not analyzed for NSCLC arm because there was insufficient data to perform the DC analysis.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | mCRPC: Isatuximab + REGN2810 | NSCLC: Isatuximab + REGN2810
Number analyzed (Participants) | 24 | 0
percentage of participants | 20.8 [8.6 to 38.9] |

ADVERSE EVENTS:
Time Frame: From Baseline up to 30 days after the last dose of study treatments (maximum duration: up to 2 years)
Description: Reported adverse events (AE) and deaths were TEAEs i.e., AE that developed, worsened, or became serious during the TEAE period (time from the first dose of study treatment up to 30 days after last dose of study treatment). Analysis was performed on all-treated population.
Arm/Group | mCRPC: Isatuximab + REGN2810 | NSCLC: Isatuximab + REGN2810
All-Cause Mortality (participants affected / at risk) | 2/24 | 2/20
Serious Adverse Events (participants affected / at risk) | 11/24 | 14/20
Other Adverse Events (participants affected / at risk) | 24/24 | 19/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | mCRPC: Isatuximab + REGN2810 (N=24) | NSCLC: Isatuximab + REGN2810 (N=20)
Atrial Fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Immune-Mediated Enterocolitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Intestinal Obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Malignant Dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Disease Progression (General disorders) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 2 (2)
Urinary Tract Infection (Infections and infestations) | 1 (1) | 0 (0)
Urosepsis (Infections and infestations) | 1 (1) | 0 (0)
Infusion Related Reaction (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Post Procedural Haematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Back Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Spinal Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Cancer Pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Malignant Pleural Effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (3) | 0 (0)
Metastases To Peritoneum (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Metastases To Spinal Cord (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Tumour Necrosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 0 (0)
Spinal Cord Compression (Nervous system disorders) | 0 (0) | 1 (1)
Hydronephrosis (Renal and urinary disorders) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Immune-Mediated Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 1 (1)
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | mCRPC: Isatuximab + REGN2810 (N=24) | NSCLC: Isatuximab + REGN2810 (N=20)
Abdominal Pain (Gastrointestinal disorders) | 2 (2) | 2 (2)
Abdominal Pain Upper (Gastrointestinal disorders) | 1 (1) | 3 (3)
Constipation (Gastrointestinal disorders) | 2 (2) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 5 (6) | 2 (2)
Nausea (Gastrointestinal disorders) | 4 (4) | 3 (3)
Stomatitis (Gastrointestinal disorders) | 2 (2) | 0 (0)
Vomiting (Gastrointestinal disorders) | 3 (5) | 2 (2)
Asthenia (General disorders) | 6 (6) | 4 (4)
Fatigue (General disorders) | 8 (8) | 3 (3)
Oedema Peripheral (General disorders) | 5 (5) | 0 (0)
Pyrexia (General disorders) | 6 (8) | 4 (4)
Bronchitis (Infections and infestations) | 0 (0) | 2 (2)
Rhinitis (Infections and infestations) | 0 (0) | 2 (2)
Upper Respiratory Tract Infection (Infections and infestations) | 3 (5) | 1 (1)
Urinary Tract Infection (Infections and infestations) | 2 (3) | 0 (0)
Infusion Related Reaction (Injury, poisoning and procedural complications) | 10 (10) | 8 (8)
Decreased Appetite (Metabolism and nutrition disorders) | 9 (9) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Back Pain (Musculoskeletal and connective tissue disorders) | 7 (8) | 1 (2)
Bone Pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 3 (4) | 0 (0)
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 3 (4) | 1 (1)
Dizziness (Nervous system disorders) | 2 (2) | 2 (3)
Hypoaesthesia (Nervous system disorders) | 2 (2) | 0 (0)
Paraesthesia (Nervous system disorders) | 0 (0) | 2 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 6 (9)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (2)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (3)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (4)
Dry Skin (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Pruritus (Skin and subcutaneous tissue disorders) | 4 (5) | 3 (3)
Deep Vein Thrombosis (Vascular disorders) | 2 (2) | 0 (0)
Hypertension (Vascular disorders) | 3 (4) | 1 (1)
Hypotension (Vascular disorders) | 2 (2) | 2 (2)

LIMITATIONS AND CAVEATS:
The study was terminated after the interim analysis of the primary endpoint. Few planned outcome measures per-protocol were not analyzed because overall efficacy results were not sufficient at the time of interim analyses of both the cohorts.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor supports publication of clinical trial results but may request that investigators temporarily delay or alter publications in order to protect proprietary information. The Sponsor may also require that the results of multicenter studies be published only in their entirety and not as individual site data.

DOCUMENTS (2):
  • Study Protocol (2019-06-11): https://cdn.clinicaltrials.gov/large-docs/19/NCT03367819/Prot_000.pdf
  • Statistical Analysis Plan (2018-12-17): https://cdn.clinicaltrials.gov/large-docs/19/NCT03367819/SAP_001.pdf